CLINICAL TRIAL: NCT02610894
Title: A mHealth Self-Management Program to Decrease Postoperative Symptom Distress in Orthopaedic Patients
Brief Title: An mHealth Self-Management Program to Decrease Postoperative Symptom Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jan Odom Forren (Other)
Responsible Party: Sponsor-Investigator, Jan Odom Forren, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-0340-P6H
Record Dates: First submitted 2015-11-09; First posted 2015-11-20 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Orthopaedic Surgery
Keywords: postoperative symptom management; symptom management; mHealth application

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth application (Experimental): Participants will be provided an iPad Mini tablet computer loaded with an mHealth application (PoCAH) to provide enhanced post-operative pain care management. The app will utilize algorithms tailored to the patient's needs and symptoms in an attempt to reduce poor outcomes related to post-operative pain management.
  Interventions: Other: mHealth application (PoCAH)
- Control Group (Active Comparator): Participants will be provided an iPad Mini tablet computer loaded with a PDF of the As usual standard discharge and care instructions for post-operative pain care management.
  Interventions: Other: As usual standard discharge and care instructions

INTERVENTIONS:
Other: mHealth application (PoCAH) — Participants will have unlimited access to the mHealth app via iPad Mini for 5 days post-operatively to aid in pain management
  Arms: mHealth application
Other: As usual standard discharge and care instructions — As usual standard discharge and care instructions are provided via iPad mini to orthopaedic ambulatory surgery patients.
  Arms: Control Group

SUMMARY:
The purposes of this study are to determine if use of the Postoperative Care at Home (PoCAH) tailored self-management program delivered via mobile technology (a mobile app) after discharge to home will result in: 1) fewer and/or less intense patient symptoms (pain, nausea and vomiting, fatigue, sore throat, constipation, sleep dysfunction); 2) enhanced patient satisfaction, perceived self-efficacy, and quality of life; 3) lower healthcare resource use (patient to healthcare provider calls; unscheduled patient appointments with healthcare providers; and hospital readmission and emergency department use). A secondary objective is to assess how easy the mobile app was to use after orthopaedic ambulatory surgery.

DETAILED DESCRIPTION:
The purposes of the single-blind randomized, controlled comparative effectiveness trial are to determine if use of the Postoperative Care at Home (PoCAH) tailored self-management program delivered via mobile technology after discharge to home will result in: 1) fewer and/or less intense patient symptoms (pain, nausea and vomiting, fatigue, sore throat, constipation, sleep dysfunction); 2) enhanced patient satisfaction, perceived self-efficacy, and quality of life; 3) lower healthcare resource use (patient to healthcare provider calls; unscheduled patient appointments with healthcare providers; and hospital readmission and emergency department use). A secondary objective is to assess the utility and effectiveness of the mHealth app after orthopaedic ambulatory surgery. This is a single-blind, two-group randomized, controlled comparative effectiveness trial stratified by knee and shoulder surgical procedures (N = 40; 20 per procedure, with half in each procedure group randomized to each treatment group) to compare the effectiveness of treatment as usual to treatment as usual combined with PoCAH. PoCAH is a theory based, patient-centered, and tailored self-management program delivered via mHealth technology to orthopaedic ambulatory surgery patients. Patients in the treatment as usual group will receive standard discharge and care instructions provided on an iPad mini. Patients in the intervention group (treatment as usual combined with PoCAH) will have access to the PoCAH app, in addition to the standard discharge and care instructions. The PoCAH app will provide the patient with additional information regarding self-management of symptoms and other consequences of surgery. Orthopaedic patients who undergo knee and shoulder ambulatory surgery will be recruited because these patients typically report more postoperative symptom distress than patients undergoing other surgical procedures. The sample will consist of 40 adults recruited from the University of Kentucky Orthopaedic Surgery and Sports Medicine Clinic in Lexington, Kentucky. After consent is obtained, all patients, regardless of grouping, will complete assessments (a Patient Diary) at enrollment (i.e., baseline), which will query/assess demographic information, health literacy, quality of life, quality of recovery and perceived self-efficacy of symptom management. Health literacy will be acquired preoperatively in the event literacy is a confounding factor in use of the app. These materials will be collected by the researcher at that time. During surgery, patients will undergo anesthesia as determined by the anesthesia provider and receive usual surgical care preoperatively and postoperatively. Medical chart data regarding the surgery will be abstracted and will include length of surgery, length of stay in the Post Anesthesia Care Unit (PACU), medications/anesthetics administered, and information regarding pain and nausea in the PACU and Phase 2 Recovery (Step-Down Unit). After surgery, data will be collected daily for 5 days from all participants (Day 1 through Day 5) via a Patient Diary. The Patient Diary will contain previously validated questionnaires that will assess Quality of Life, Quality of Recovery, and postoperative symptoms. The Patient Diary will be completed in the patients' homes while they recover. The investigators will call the patients at home on Day 2 to facilitate data collection. At the conclusion of the study (Day 5), participants in the intervention group will evaluate the utility and effectiveness of the PoCAH app. The iPad minis and Patient Diaries will be returned to the research staff when the patient attends the physician's office on the first office visit at 5 days post-surgery. Because the course of post discharge symptoms extends past 5 days, phone interviews at 2 weeks and 4 weeks are included to better describe the recovery trajectory and outcomes for operative patients.

ELIGIBILITY:
Inclusion Criteria:

1. individuals of either gender and any ethnicity;
2. general and regional anesthesia for a shoulder or knee procedure;
3. surgery scheduled at the UK Center for Advanced Surgery (CAS);
4. age greater than or equal to 18

Exclusion Criteria:

1. chronic pain or nausea unrelated to surgery;
2. inability to speak or read English;
3. diagnosed cognitive dysfunction;
4. disabilities that limit the capability to manipulate the mHealth device (iPad mini);
5. visual impairment;
6. unscheduled admission after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

PRIMARY OUTCOMES:
Change in perceived pain | baseline, day 1, day 2, day 3, day 4, day 5, day 14, day 28
  Participants will be asked on multiple occasions (pre-operative assessment,day 1, day 2, day 3, day 4, day 5, day 14 and day 28) to rate their pain on a scale of 0-10. Zero would indicate no pain and 10 would represent the worst pain imaginable. Data will be presented as the change in perceived pain over the course of 28 days.

SECONDARY OUTCOMES:
Change in perceived self efficacy | baseline, day 1, day 5, day 14, day 28
  Instrument specifically designed to measure perceived self-efficacy to manage postoperative symptoms and conditions of postoperative care. Participants will be asked a series of questions with scores ranging from 0-10 where 10 represents absolute self confidence in a task and 0 represents no confidence in a task. Data will be presented as the change in self-efficacy over the course of 28 days. Data will be collected at the following time points: preoperative assessment, Day 1, Day 5, day 14,and day 28.
Change in quality of life | baseline, day 1, day 5, day 14, day 28
  The European Quality of Life Survey includes questions addressing the following five categories: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Participants will be asked to answer the questions with the following five responses: no problems, slight problems, moderate problems, severe problems, and extreme. Answers are scored on a 1-5 scale and combined into a 5 digit number conveying the participants overall quality of life. Data will be presented as the change in quality of life over the course of 28 days. Data will be collected at the following time points: preoperative assessment, Day 1, Day 5, day 14,and day 28.
Change in postoperative heath status | preoperative assessment, Day 1, Day 5, day 14,and day 28.
  The Quality of Recovery Patient Survey (QoR-15) is a 15 question survey that measures early postoperative health status. Each question is answered on a scale of 0-10 were 10 is a very positive answer and zero is the worst possible scenario. Data will be presented as the change in postoperative health status over the course of 28 days. The assessment will take place preoperative assessment, Day 1, Day 5, day 14,and day 28.
Change in postoperative health status | preoperative assessment, Day 1, Day 5, day 14,and day 28.
  The Swedish Quality of Recovery Patient Survey (QoR-40) is a 40 question survey that measures early postoperative health status. Each question is answered on a scale of 0-10 were 10 is a very positive answer and zero is the worst possible scenario. Data will be presented as the change in postoperative health status over the course of 28 days. The assessment will take place preoperative assessment, Day 1, Day 5, day 14,and day 28.
Healthcare resource use | 28 days
  Number of patient to healthcare provider calls, unscheduled patient appointment with healthcare providers, hospital readmissions, emergency department visits. Data will be collected through a medical record search and presented as the total count of healthcare resources used per group in 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Odom Forren, PhD, RN, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Orthopaedic Surgery and Sports Medicine Clinic, Lexington, Kentucky, United States